CLINICAL TRIAL: NCT01499654
Title: Feasibility of Half-Dose Radiopharmaceutical Administration Utilizing Wide-Beam Reconstruction
Brief Title: Half-Dose Radiopharmaceutical in Wide Beam Reconstruction
Acronym: REGA-1102
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Edwin Wu (Other)
Collaborators: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Edwin Wu, Associate Professor of Medicine and Radiology, Northwestern University
Organization: Northwestern University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STU53243
Record Dates: First submitted 2011-12-19; First posted 2011-12-26 (Estimated); Results first posted 2016-02-24 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-01

CONDITIONS: Myocardial Infarction; Ischemic Heart Disease
Keywords: SPECT MPI; Tomography, Emission-Computed, Single-Photon; Wide Beam Reconstruction
MeSH Terms: conditions — Myocardial Infarction; Myocardial Ischemia | interventions — Technetium Tc 99m Sestamibi; Technetium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Half-dose radiotracer administration (Experimental): For this study, researchers would like to administer half of the radiotracer, obtain resting images, administer the remainder of the radiotracer and obtain a second set of resting images. Subjects will be given the same amount of radioactive material that would normally be given for this test; however, it will be administered in two ½ doses.
  Interventions: Drug: Half-dose of the Tc99-m sestamibi (Cardiolite)

INTERVENTIONS:
Drug: Half-dose of the Tc99-m sestamibi (Cardiolite) — Researchers will administer half of the radiotracer (Cardiolite), obtain resting images, administer the remainder of the radiotracer and obtain a second set of resting images. Subjects will be given the same amount of radioactive material that would normally be given for this test; however, it will be administered in two ½ doses.
  Other Names: technetium (Tc-99m) sestamibi, Cardiolite

SUMMARY:
This study is recruiting patients already scheduled for a single photon emission computed tomography myocardial perfusion imaging (SPECT-MPI) test. SPECT-MPI is a nuclear imaging technique that uses a radioactive substance, or radiotracer, and special equipment to create three-dimensional (3D) images of the heart. Radiotracer is a radioactive dye that will make the structures of the heart visible and is routinely used to view blood flow in the heart, scan for damaged heart tissue, or assess heart function.

For a routine SPECT-MPI test, the radiotracer is given in one dose at the beginning of the test, followed by taking resting images of the heart. For this study, researchers would like to administer half of the radiotracer, obtain resting images, administer the remainder of the radiotracer and obtain a second set of resting images. Participants will receive the same amount of radioactive material that would normally be given for this test; however, it will be administered in two half-doses. Participation in this study will add about 30 minutes to the time it takes to complete the routine test. The investigators expect to enroll about 160 subjects in this study at Northwestern.

DETAILED DESCRIPTION:
Subjects in this study will proceed to the nuclear cardiology laboratory for their scheduled nuclear stress test. After informed consent is obtained, the study doctor or research staff member will ask detailed questions about the subject's current health, medications and medical history, and the subject's medical chart will be reviewed including results of any previous nuclear images.

For the test, a small catheter (tube) will be placed in a vein in the subject's arm to administer the radioactive imaging agent, Tc-99m sestamibi. Subjects will be given half (1/2) of the normal Tc-99m sestamibi dose and then the study staff will obtain resting images pictures of the heart. After this set of images, the subject will be given the remaining half of the radioactive imaging agent followed by a second set of images.

After this, the subject will then undergo the stress portion of the test in the usual manner as prescribed by the referring physician.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 years
* Undergoing nuclear stress testing
* History of myocardial infarction, cardiomyopathy, heart failure or prior nuclear studies with resting perfusion defects

Exclusion Criteria:

* Unwilling or unable to undergo an additional resting SPECT acquisition
* Clinical contraindications to nuclear stress testing including acute myocardial infarction

  * For patients undergoing exercise treadmill stress testing:
* Left bundle branch block or artificial ventricular pacemaker

  * For patients undergoing regadenoson (Lexiscan) stress testing:
* Moderate to severe chronic obstructive pulmonary disease or asthma, second- or third degree atrioventricular block or sinus node disease (unless patients have a functioning artificial pacemaker), known hypersensitivity to aminophylline or adenosine
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2011-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edwin Wu, M.D., FACC, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Prospectively enroll patients with history of severe myocardial infarction, cardiomyopathy, heart failure or prior nuclear scans with resting perfusion defects. Patients were approached in the nuclear stress lab prior to scheduled stress test. Recruitment period was between 3/20/2012 and 2/14/2014.
Groups:
- Study Group: Entire cohort
Period: Overall Study
Arm/Group | Study Group
Started | 64
Completed | 64
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Study Group
Number analyzed (Participants) | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 48
Height [Mean (Standard Deviation); unit: inches] | 68.0 (4.1)
Weight [Mean (Standard Deviation); unit: pounds] | 198.4 (40.0)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 30.2 (6.0)
Indications for stress test [Number; unit: participants]
  Chest pain | 16
  Dyspnea | 9
  Prior Myocardial Infarct | 7
  Prior Coronary Disease | 18
  Cardiomyopathy | 5
  CHF | 6
  Prior CABG | 8
  Prior PCI | 5
  Other | 9
History [Number; unit: participants]
  Hypertension | 58
  Hypercholesterolemia | 52
  Tobacco smoking (prior or current) | 24
  Diabetes mellitus | 21
  Family history of CAD | 19
  Prior Myocardial Infarct | 28
  Coronary artery disease | 46
  Coronary artery bypass surgery | 27
Previous nuclear stress [Number; unit: participants] | 39
Medications [Number; unit: participants]
  ACE inhibitors/ARB | 33
  Beta-blockers | 56
  Ca-channel blockers | 19
  Aspirin | 51
  Anti-platelet | 21
  Statin | 53
  Nitrates | 11
  Diuretic | 24

OUTCOME MEASURES:

1. Primary Outcome: Sum Rest Score
Description: Left ventricular myocardium was divided into standardized 17-segments with 6 equiangular segments in the basal region, 6 equiangular segments in the mid region, 4 equiangular segments in the apical regions, and 1 region in the apex (Cerqueira MD, et al., J Nucl Cardiol 2002;9:240-5). Each segment was scored on a scale from 0 to 4 to indicate the severity of the perfusion defect (0=no perfusion defect; 1=mild perfusion defect; 2=moderate perfusion defect; 3=severe perfusion defect; and 4=absent perfusion). The scores over 17 segments were summed to report the Sum Rest Score (SRS), ie. the greater the SRS, the larger the perfusion defect.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Half-dose WBR: Half-dose Tc-99m sestamibi reconstructed using wide beam reconstruction (WBR)
- Half-dose FBP: Half-dose Tc-99m sestamibi reconstructed using filtered back projection (FBP)
- Full-dose FBP: Full-dose Tc-99m sestamibi reconstructed using filtered back projection (FBP)
Arm/Group | Half-dose WBR | Half-dose FBP | Full-dose FBP
Number analyzed (Participants) | 64 | 64 | 64
units on a scale | 8.1 (5.9) | 6.7 (5.1) | 6.5 (6.1)
Statistical Analysis 1: Comparison: Half-dose WBR vs Full-dose FBP; Test type: Superiority or Other; p = 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Half-dose FBP vs Full-dose FBP; Test type: Superiority or Other; p = 0.67, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Image Quality Score
Description: Each reconstructed image was subjectively scored by the expert readers to determine the overall image quality. The Image Quality Score of the reconstructed images were graded on a 4-point scale. (1=Poor; 2=Fair; 3=Good; and 4=Excellent).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Half-dose WBR | Half-dose FBP | Full-dose FBP
Number analyzed (Participants) | 64 | 64 | 64
units on a scale | 2.3 (0.8) | 2.6 (0.6) | 3.0 (0.7)
Statistical Analysis 1: Comparison: Half-dose WBR vs Full-dose FBP; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Half-dose FBP vs Full-dose FBP; Test type: Superiority or Other; p = 0.002, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Diagnostic Confidence Score
Description: Each reconstructed image was subjectively scored by the expert readers to determine the expert reader's diagnostic confidence in scoring and interpreting the perfusion scores. The Diagnostic Confidence Score of the reconstructed images were graded on a 4-point scale. (1=Poor; 2=Fair; 3=Good; and 4=Excellent).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Half-dose WBR | Half-dose FBP | Full-dose FBP
Number analyzed (Participants) | 64 | 64 | 64
units on a scale | 2.5 (0.8) | 2.7 (0.9) | 3.0 (0.8)
Statistical Analysis 1: Comparison: Half-dose WBR vs Full-dose FBP; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Half-dose FBP vs Full-dose FBP; Test type: Superiority or Other; p = 0.08, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Segments With Resting Perfusion Defect
Description: Left ventricular myocardium was divided into standardized 17-segments with 6 equiangular segments in the basal region, 6 equiangular segments in the mid region, 4 equiangular segments in the apical regions, and 1 region in the apex (Cerqueira MD, et al., J Nucl Cardiol 2002;9:240-5). Each segment was scored on a scale from 0 to 4 to indicate the severity of the perfusion defect (0=no perfusion defect; 1=mild perfusion defect; 2=moderate perfusion defect; 3=severe perfusion defect; and 4=absent perfusion). The number of segments with a score of 1 or greater were summed to obtain the number of segments with a resting perfusion defect.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: segments
Arm/Group | Half-dose WBR | Half-dose FBP | Full-dose FBP
Number analyzed (Participants) | 64 | 64 | 64
segments | 4.6 (2.4) | 4.0 (2.2) | 3.8 (2.6)
Statistical Analysis 1: Comparison: Half-dose WBR vs Full-dose FBP; Test type: Superiority or Other; p = 0.006, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Half-dose FBP vs Full-dose FBP; Test type: Superiority or Other; p = 0.44, Wilcoxon (Mann-Whitney)

5. Post Hoc Outcome: Resting Full-Tracer Dose
Description: Amount of the standard, clinically-accepted, full-dose Tc-99m sestamibi dose administered
Time Frame: Baseline
Population: Entire Cohort
Measure: Mean (Standard Deviation); unit: millicurie
Arm/Group | Study Group
Number analyzed (Participants) | 64
millicurie | 9.08 (0.46)

6. Post Hoc Outcome: Injection and Scan Times
Description: Time in minutes between doses of resting Tc-99m sestamibi doses and image scanning.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Injection 1 to Scan 1: Time in minutes between the first 1/2 dose injection and the first scan
- Injection 2 to Scan 2: Time in minutes between the second 1/2 dose injection and the second scan.
- Injection 1 to Injection 2: Time in minutes between the first 1/2 dose injection and the second 1/2 dose injection
Arm/Group | Injection 1 to Scan 1 | Injection 2 to Scan 2 | Injection 1 to Injection 2
Number analyzed (Participants) | 64 | 64 | 64
minutes | 30.0 (5.4) | 33.1 (13.1) | 56.7 (8.2)

ADVERSE EVENTS:
Time Frame: Adverse events were only collected during the time frame of the imaging study, ie. between the first 1/2 dose injection and the second imaging scan (Reference Outcome Measures, post-hoc analysis "Injection and Scan Times").
Description: Adverse events for this imaging study would include mis-administration of a tracer dose or errors in acquiring images that would result in an inability to interpret and report the clinical imaging study to the referring physician.
Groups:
- Study Group: Entire cohort for the study
Arm/Group | Study Group
Serious Adverse Events (participants affected / at risk) | 0/64
Other Adverse Events (participants affected / at risk) | 0/64

LIMITATIONS AND CAVEATS:
Early termination of study lead to a small numbers of subjects analyzed. Technical problems in WBR processing settings including acquisition matrix sizes and/or number of iterations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No